CLINICAL TRIAL: NCT02261636
Title: Induction and Maintenance of Remission With Pentasa as Ulcerative Colitis Treatment
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000157
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2019-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pentasa: Treatment according to standard clinical practice.
  Interventions: Drug: mesalazine

INTERVENTIONS:
Drug: mesalazine
  Other Names: Pentasa

SUMMARY:
For both induction of remission and in maintenance of remission, different doses and treatment durations are used in practice. The aim of this study is to assess how mesalazine is used in clinical practice, at which doses and for how long and how these differences impact the patient disease state and work productivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate active ulcerative colitis with disease extension beyond the rectum (≥ 10 cm) who will receive oral Pentasa treatment (Compact sachets and/or tablets) for the treatment of the current active episode or in whom on oral Pentasa maintenance treatment induction of remission treatment will be initiated by dose escalation. Treatment combined with Pentasa enema (1g/100ml) is allowed.
* Informed consent

Exclusion Criteria:

* Patients receiving treatment with one or more of the following: locally acting steroids (e.g. budesonide, beclomethasone), systemic steroids, immunosuppressants (e.g. thiopurines), biologicals (e.g. anti-Tumor Necrosis Factor-alpha)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patient clinics in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Time to dose reduction | From Day 1 up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Gelre Ziekenhuizen (there may be other sites in this country), Zutphen, Netherlands

REFERENCES:
- [Result] West R, Russel M, Bodelier A, Kuijvenhoven J, Bruin K, Jansen J, Van der Meulen A, Keulen E, Wolters L, Ouwendijk R, Bezemer G, Koussoulas V, Tang T, Van Dobbenburgh A, Van Nistelrooy M, Minderhoud I, Vandebosch S, Lubbinge H. Lower Risk of Recurrence with a Higher Induction Dose of Mesalazine and Longer Duration of Treatment in Ulcerative Colitis: Results from the Dutch, Non-Interventional, IMPACT Study. J Gastrointestin Liver Dis. 2022 Mar 19;31(1):18-24. doi: 10.15403/jgld-3927. PMID 35306553